CLINICAL TRIAL: NCT07317570
Title: A Randomized, Single-Blind Controlled Trial Investigating the Effect of Body Awareness Therapy on Pain, Functional Outcomes, and Psychosocial Parameters in Adults With Temporomandibular Joint Disorders
Brief Title: The Effect of Body Awareness Therapy on Pain, Function and Psychosocial Parameters in Temporomandibular Joint Disorders
Acronym: BAT-TMJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Seda Karaca, Principal Investigator, Doctor Lecturer, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/457
Record Dates: First submitted 2025-12-07; First posted 2026-01-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Awareness Therapy (BAT) (Experimental): Participants will receive Body Awareness Therapy
  Interventions: Behavioral: Body Awareness Therapy; Other: Standard Physiotherapy
- Standard Physiotherapy (Other): Participants will receive standard physiotherapy
  Interventions: Other: Standard Physiotherapy

INTERVENTIONS:
Behavioral: Body Awareness Therapy — Body Awareness Therapy
  Arms: Body Awareness Therapy (BAT)
Other: Standard Physiotherapy — Standard Physiotherapy

SUMMARY:
This randomized, single-blind controlled trial aims to investigate the effectiveness of Body Awareness Therapy (BAT) on pain, functional limitations, and psychosocial outcomes in individuals with temporomandibular joint disorders (TMD). TMD is characterized by orofacial pain, impaired jaw function, and increased psychosocial burden, yet current physiotherapy approaches may not fully address the biopsychosocial mechanisms underlying these symptoms. BAT is a structured mind-body physiotherapy intervention designed to improve postural awareness, interoceptive sensitivity, breathing regulation, and movement control.

In this study, participants will be randomly assigned to either BAT or a standard physiotherapy control intervention for a defined treatment period. Primary outcomes will include pain intensity and jaw functional limitations, while secondary outcomes will assess body awareness, anxiety, stress, and quality of life. Evaluations will be conducted at baseline and post-intervention. The findings of this trial may provide evidence for integrating biopsychosocial and awareness-based physiotherapy into TMD rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years. Diagnosed with Temporomandibular Joint Disorders (TMD) according to the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).

Experiencing orofacial pain or jaw functional limitation for at least the past 3 months.

Ability to understand and follow verbal instructions required for Body Awareness Therapy sessions.

Willingness to participate in the study and to attend all assessment and intervention sessions.

Providing written informed consent.

Exclusion Criteria:

History of jaw trauma, fracture, or surgery within the past 6 months. Presence of systemic rheumatologic or inflammatory disorders (e.g., rheumatoid arthritis, ankylosing spondylitis) that may affect TMJ function.

Neurological or psychiatric conditions that could interfere with participation or outcome assessments (e.g., major psychiatric disorder, cognitive impairment).

Severe dental or orthodontic conditions requiring immediate treatment (e.g., acute infection, ongoing orthodontic procedures).

Use of occlusal splints, bite guards, or other TMJ-related interventions initiated within the past 3 months.

Participation in any other physiotherapy or exercise program targeting the jaw, cervical spine, or posture during the study period.

Pregnancy, due to potential changes in joint laxity and pain perception. Current use of medications affecting neuromuscular or pain responses, such as muscle relaxants, corticosteroids, or neuropathic pain medications (unless dose has been stable for 3 months).

Any contraindication to performing light-to-moderate physical activity or awareness-based exercises.

Inability to attend scheduled therapy sessions or complete study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Jaw Functional Limitation Scale (JFLS) | Baseline, post-intervention (8 weeks)
  Jaw functional limitation assessed by the Jaw Functional Limitation Scale (JFLS). Change in jaw-related functional limitation measured using the Jaw Functional Limitation Scale (JFLS), a validated self-report questionnaire assessing limitations in mastication, jaw mobility, and verbal communication. The total score ranges from 0 to 200, with higher scores indicating greater functional limitation (worse outcome).
Hospital Anxiety and Depression Scale | Baseline, post-intervention (8 weeks)
  Change in anxiety and depression levels measured using the Hospital Anxiety and Depression Scale (HADS), a validated 14-item self-report questionnaire. The anxiety (HADS-A) and depression (HADS-D) subscales are each scored from 0 to 21, with higher scores indicating greater symptom severity (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Guneysu Physical Therapy and Rehabilitation School, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and institutional ethical restrictions. The study involves sensitive health information, and the ethics committee approval covers data use only within the scope of this research. De-identified datasets cannot be made publicly available to ensure participant confidentiality is maintained.